CLINICAL TRIAL: NCT06896435
Title: Smart-Phone Safety Behavior Fading Intervention for Appearance Concerns
Brief Title: Smart-Phone Safety Behavior Fading Intervention for Appearance Concerns (Open ARSB Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Jesse Cougle, Principal Investigator, Florida State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00005977
Record Dates: First submitted 2025-03-20; First posted 2025-03-26 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Body Dysmorphic Disorder; Social Anxiety Disorder; Eating Disorders
Keywords: appearance concerns; safety behavior
MeSH Terms: conditions — Body Dysmorphic Disorders; Phobia, Social; Feeding and Eating Disorders

STUDY DESIGN:
Intervention Model Description: Participants are randomized to one of two conditions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Safety Behavior Fading (Experimental): Individuals randomly assigned to the safety behavior fading condition will receive instructions to decrease or eliminate their endorsed appearance-related safety behaviors. In addition, they will receive daily reminders via text message to decrease these behaviors, along with a safety behavior monitoring checklist in which the participant indicates the extent to which they engaged in each safety behavior over the previous day.
  Interventions: Behavioral: Safety Behavior Fading for Appearance Concerns
- Relaxing Video (Active Comparator): Individuals randomly assigned to the relaxing video condition will receive a total of 4 videos over the course of a month (1 video per week, 15 minutes each) wherein participants will be invited to close their eyes and focus their attention on the present moment while listening to relaxing piano music and songbirds.
  Interventions: Behavioral: Relaxing Video

INTERVENTIONS:
Behavioral: Safety Behavior Fading for Appearance Concerns — Participants are asked to reduce or eliminate safety behaviors via text message reminders and checklists to monitor progress.
  Arms: Safety Behavior Fading
Behavioral: Relaxing Video — Participants are asked to view weekly videos lasting 15 minutes each to engage in relaxation exercises.
  Arms: Relaxing Video

SUMMARY:
The current study aims to explore the efficacy of a text message based safety behavior fading intervention compared to a relaxing video intervention for appearance concerns.

DETAILED DESCRIPTION:
Description: Appearance-related safety behavior fading intervention procedures will follow methodology previously used in the Cougle Lab. The safety behavior fading intervention is designed to target a decrease or elimination of appearance-related safety behaviors. Individuals randomly assigned to the safety behavior fading condition will receive instructions to decrease or eliminate their endorsed appearance-related safety behaviors. In addition, they will receive daily reminders via text message to decrease these behaviors, along with a safety behavior monitoring checklist in which the participant indicates the extent to which they decreased and/or eliminated each safety behavior over the previous day. The daily reminder will include the following language: "Hi! This is a friendly reminder to avoid using your checklist behaviors. Please tap the link below to access today's checklist: [link to checklist]." Text messages will be delivered using EZtexting a text messaging platform used for research and marketing. Note that no identifying information will be included in this platform. Each participants phone number will be accompanied with a anonymized ID code. Individuals randomly assigned to the relaxing video condition will receive a total of 4 videos over the course of a month (1 video per week, 15 minutes each) wherein participants will be invited to close their eyes and focus their attention on the present moment while listening to relaxing piano music and songbirds.

ELIGIBILITY:
Inclusion Criteria:

* Seeking treatment for appearance concerns

Exclusion Criteria:

* Currently receiving treatment (therapy, counseling, etc.) for anxiety, depression, eating disorder, or body image/appearance concerns
* If applicable, unstable psychiatric medication usage any time over the past 4 weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-09-08 (Actual); Study Completion 2025-09-08 (Actual)

PRIMARY OUTCOMES:
The Social Appearance Anxiety Scale (SAAS; Hart et al., 2008) | Day 0, Day 28, Day 56
  Self-report scale that measures appearance anxiety symptoms. Scores range from 16 to 80 with higher scores indicating higher levels of appearance concerns.
Social Phobia Inventory (SPIN; Connor et al., 2000) | Day 0, Day 28, Day 56
  Self-report scale that measures social anxiety symptoms. Scores range from 0 to 68 with higher scores indicating higher levels of social anxiety.
Credibility and Expectancy Questionnaire (Devilly & Borkovec, 2000). | Day 0
  Self-report scale for measuring treatment expectancy and rationale credibility for use in clinical outcome studies. Three items are rated on a 0-10 scale and one item is rated on a 0-100 scale with higher scores meaning greater expectancy and credibility.
Eating Disorder Inventory (EDI; Garner et al., 1983). | Day 0, Day 28, Day 56
  Self-report scale for measuring drive for thinness, bulimia, and body dissatisfaction for use in clinical outcome studies. Each item is rated on a 0-5 scale with a total score range of 0-125 with higher scores indicating greater drive for thinness, bulimia, and body dissatisfaction.
Appearance Behaviors Checklist past-week version (author constructed) | Day 0, Day 28, Day 56
  Self-report scale used to measure frequency of engaging in appearance-related safety behaviors. This scale will be used as a manipulation check. Each item is rated on a 0 to 10 scale. Total scores range from 0 to 130 with higher scores indicating greater engagement in appearance-related safety behaviors

SECONDARY OUTCOMES:
Distress Intolerance Index (McHugh & Otto, 2012) | Day 0, Day 28, Day 56
  Self-report scale for measuring tolerance to distress for use in clinical outcome studies. Each item is rated on a 0-4 scale with a total score range of 0-40 with higher scores indicating greater intolerance of distress.
Frost Multidimensional Perfectionism Scale-Concerns over mistakes subscale (Frost et al., 1990) | Day 0, Day 28, Day 56
  Self-report scale for measuring concerns for making mistakes for use in clinical outcome studies. Each item is rated on a 0-4 scale with a total score range of 0-36 with higher scores indicating greater concerns for making mistakes.
Center for Epidemiologic Studies Depression Scale-10 (CESD; Andreson, 1994) | Day 0, Day 28, Day 56
  Self-report measure of depression symptom severity. Each item is rated on a 0 to 3 scale. Total scores range from 0 to 30 with higher scores indicating greater depression severity.

CONTACTS AND LOCATIONS:
Overall Officials: Jesse Cougle, Doctor of Philosophy, Study Director — Florida State University
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No